CLINICAL TRIAL: NCT05327608
Title: Time Restricted Eating for Patients With HER2- Negative Breast Cancer Receiving Neoadjuvant Chemotherapy
Brief Title: Neoadjuvant Breast Cancer Time Restricted Eating
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 21D.625; JT 16674 (Other: JeffTrial Number)
Record Dates: First submitted 2021-12-13; First posted 2022-04-14 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Breast Ductal Carcinoma in Situ; HER2 Negative Breast Carcinoma; Hormone Receptor Positive Breast Carcinoma; Invasive Breast Carcinoma
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Time Restricted Eating) (Experimental): This is a single arm, non-randomized trial. All participants will undergo TRE for 16 weeks while receiving NCT. For patients requiring NCT longer than 16 weeks, they can continue TRE however this will not be included in the main adherence calculations.
  Interventions: Other: Time Restricted Eating

INTERVENTIONS:
Other: Time Restricted Eating — Undergo intermittent fasting
  Other Names: Short-term Intermittent Fasting

SUMMARY:
A phase II study to evaluate an innovative approach of following time restricted eating (TRE) in patients with HER2- negative breast cancer who will start neoadjuvant chemotherapy (NCT) for a new diagnosis of stage I-III breast cancer. Participants at baseline will have a body mass index (BMI) of (25-40) and engage in a TRE 16:8 schedule which includes 16 hours of fasting and 8 hours of eating. Patients will continue TRE for 16 weeks while receiving NCT. For patients who report at the time of the 2-3 week clinic visit that they are finding it challenging to adhere to the 16:8 TRE, instructions will be provided about alternative measures such as changing the time of the day they fast, dietary modifications and finally changing to a 14:10 schedule if other measures fail. For patients requiring NCT for longer than 16 weeks, they will be encouraged to continue TRE. Adherence calculation for the primary endpoint will include data for the first 16 weeks, and then monitored separately for any additional optional fasting beyond the first 16 weeks. Adherence to TRE will be self-reported by patients daily through electronic surveys through RedCap and approximately every 2-3 weeks (+/- 5 days) by the research team during their clinic visit.

DETAILED DESCRIPTION:
Primary objective:

1. To evaluate the proportion of patients that can adhere to Time Restricted Eating (TRE) in patients with HER2 negative breast cancer who receive neoadjuvant chemotherapy (NCT) for a new diagnosis of stage I-III breast cancer.

Secondary objectives:

1. To evaluate the pathologic complete response (pCR) rate of TRE in patients with HER2 negative breast cancer who receive NCT for a new diagnosis of stage I-III breast cancer
2. To evaluate the effect of TRE on weight management (prevention of weight gain), measured by BMI and waist circumference, in patients who are undergoing NCT.
3. To evaluate the percent of patients who develop CTCAE version 5.0 grade 3 or 4 toxicities
4. To evaluate the differences in the pCR rate among breast cancer patients within different race/ethnic groups, African American vs. Non-Hispanic White (AA vs NHW), and based on baseline social determinants of health when undergoing NCT
5. To evaluate if study intervention acceptability, adherence, and engagement differ by race (AA vs NHW) and based on baseline social determinants of health.
6. To evaluate if percent of patients with CTCAE version 5.0 grade 3 or 4 toxicities differ by race (AA vs NHW) and based on baseline social determinants of health.

Exploratory objectives:

1. To monitor changes in the following inflammatory markers in patients undergoing neoadjuvant chemotherapy with TRE: fasting glucose, hemoglobin A1c, insulin, C-peptide, CRP, leptin, adiponectin,IGF-1, IL-6, TNF-α, and free fatty acids and lipids
2. To measure changes in markers involved in metabolic and lipogenic signaling pathways, immune modulation, and autophagy in adipocytes, tumor cells, and surrounding immune cells by Reverse-Phase Protein microarrays (RPPA) analysis. For this analysis we will use on tissue from baseline diagnostic tissue biopsies and post TRE plus neoadjuvant chemotherapy surgical tissue resection, when available

ELIGIBILITY:
Inclusion Criterion

Individuals must meet all of the following inclusion criteria in order to be eligible to participate in the study:

1. Patient must be ≥ 18 years of age at time of consent and must be able to understand and provide informed consent.
2. BMI 25-40 at time of enrollment.
3. Patients must have an ECOG performance status of 0 or 1.
4. Patient must have a recent diagnosis of histologically confirmed primary invasive breast carcinoma.

   1. Multifocal or contralateral DCIS or invasive breast cancers are allowed if the breast cancers meet the same eligibility criteria for ER/PR and HER2.
   2. Oligometastatic disease is allowed if treating physician recommends standard neoadjuvant chemotherapy.
5. Tumor status must be HER2 negative per ASCO/CAP guidelines (determined by local testing).
6. Patients must have clinical stage I-III (utilizing TNM criterion) at diagnosis.
7. Clinical T size must be ≥ 1.5cm if there is no radiographic or clinical evidence of axillary lymph node involvement. Any size tumor is allowed if axillary lymph nodes appear to be involved.
8. Patient must be willing and able (have no contraindication) to receive recommended standard neoadjuvant therapy consisting of at least 16 weeks of planned neoadjuvant chemotherapy.

   a. Acceptable regimen includes doxorubicin and cytoxan followed by a taxane The schedule will be determined by treating physician. Carboplatin and pembrolizumab can also be added to the neoadjuvant chemotherapy regimen if determined to be appropriate by treating physician.
9. Patients must have organ and marrow function adequate for initiating neoadjuvant chemotherapy as determined by their treating physician.
10. Patient must be willing and able (have no contraindication) to participate in TRE consisting of 16 weeks
11. Women of childbearing potential and sexually active males must use accepted and effective method(s) of contraception or abstain from sexual intercourse for the duration of their participation in the study and for 6 months after the last study intervention.
12. Patient must have a personal email address, an internet-capable device, and the ability/ willingness to read and reply to email every day for the duration of the study.

Exclusion Criteria

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Clinical T4 and/or N3 disease, including inflammatory breast cancer.
2. Any prior treatment for the current breast cancer diagnosis, including surgery, chemotherapy, radiation, or experimental therapy.
3. Women must not be pregnant or breast-feeding due to the potential harm to an unborn fetus and possible risk for adverse events in nursing infants with the treatment regimens being used. Patients must also not expect to conceive from the time of registration, while on study treatment, and until at least 6 months after the last study intervention.
4. Patients with type 1 diabetes, or type 2 diabetes treated with insulin.
5. Patients with a history of eating disorder or taking weight loss medications
6. Patients who actively smoke
7. Patients who work night shifts or on a rotating shift schedule.
8. Patients must not have impaired decision-making capacity.
9. Patients who are not English speaking as study staff is only able to provide the study intervention measurement tool.
10. Patients that are >2 weeks into starting neoadjuvant chemotherapy regimen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2022-07-28 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
1. Proportion of patients who can adhere to time restricted eating (TRE) >= 70% of days | While undergoing neoadjuvant chemotherapy
  A patient's adherence will be measured as the percent (%) of days where a patient reports on the survey that they were able to complete at least 14 or more hours of fasting per 24 hours (each day) during 16 weeks (112 days) of neoadjuvant chemotherapy. A patient will be considered adherent to TRE if percent (%) of days where a patient reports on the survey that they were able to complete at least 14 or more hours of fasting per 24 hours (each day) during 16 weeks is 70% or higher. For patients who complete < 16 weeks of chemotherapy from the date of starting TRE, adherence will be computed based on number of days of chemotherapy cycles received. If the proportion of days with confirmed TRE adherence is 70% or greater, then the patient is considered to have achieved overall TRE adherence.

SECONDARY OUTCOMES:
Pathologic complete response (pCR) rate | 4 months
  Will be estimated with corresponding the exact binomial 90% confidence intervals.
To measure the percent of patients who maintain or have a reduced BMI and waist circumference after TRE and neoadjuvant chemotherapy. | 4 months
  percent of patients who maintain or have a reduced BMI and waist circumference after TRE and neoadjuvant chemotherapy.
To measure the percent of patients who develop CTCAE (v5.0) grade 3 of 4 toxicities | 4 months
  percent of patients who develop CTCAE (v5.0) grade 3 of 4 toxicities
To compare pCR rate among African American vs. Non-Hispanic White breast cancer patients and based on social determinants of health when undergoing TRE plus neoadjuvant chemotherapy. | 4 months
  pCR rate among African American vs. Non-Hispanic White breast cancer
To measure the acceptability, adherence, and engagement of TRE among African American vs. Non-Hispanic White breast cancer patients and based on social determinants of health when undergoing neoadjuvant chemotherapy. | 4 months
  The acceptability, adherence and engagement of TRE among African American vs. Non-Hispanic white breast cancer patients will be measured by the percent (%) of days where a patient reports on the survey that they were able to complete at least 14 days or more hours of fasting per 24 hours ( each day) during 16 weeks ( 112 days) of neoadjuvant chemotherapy.
To evaluate if percent of patients with CTCAE (v5.0) grade 3 or 4 toxicities differs among African American vs. Non-Hispanic White breast cancer patients and based on social determinants of health when undergoing TRE plus neoadjuvant chemotherapy. | 4 months
  percent of patients with CTCAE (v5.0) grade 3 or 4 toxicities differs among African American vs. Non-Hispanic White breast cancer patients and based on social determinants of health when undergoing TRE plus neoadjuvant chemotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No